CLINICAL TRIAL: NCT04463394
Title: The Hemodynamic Effects of Vasopressin in Patients With Fontan Physiology
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manchula Navaratnam, Clinical Associate Professor, Anesthesiology, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 56875
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypotension; Fontan Physiology
MeSH Terms: conditions — Hypotension | interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: Using Minimal Sample size estimation based on the primary outcome (PVR/SVR ratio) based on paired means for decreases in PVR/SVR ratio after vasopressin administration from a prior study at our institution. We calculated a minimum sample size of 28 for a power of 0.8 and and 0.05 significant difference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vasopressin (Experimental): Participants undergoing cardiac catheterization
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Vasopressin administered intravenously

SUMMARY:
The goal of this study is to evaluate if vasopressin can elevate systemic arterial blood pressures without having a significant effect on pulmonary arterial pressures. Because patients who have undergone Fontan procedures rely on low pressures across the pulmonary vascular bed to maintain cardiac output, vasoactive agents that concomitantly increase systemic and pulmonary pressures may have a deleterious effect in this specific patient population.

Hypothesis: In patients with Fontan physiology, vasopressin will increase systemic BP by 20% above baseline, without increasing the transpulmonary gradient.

DETAILED DESCRIPTION:
Patients with Fontan physiology are at increased risk of developing hypotension during periods of illness or with anesthesia. These patients have changes in venous capacitance, compliance, and venomotor tone. When hypotension occurs, the approach to management requires a careful understanding of these changes and the selection of appropriate, efficacious vasoactive agents. Vasoconstrictive medications are frequently used to treat hypotension when patients are refractory to fluid resuscitation. However, most of these medications have an effect on both the systemic and pulmonary circulations, raising the vascular pressures of both circuits. However, these patients often do not tolerate abrupt increases in pulmonary arterial pressures or vascular resistance, and a low transpulmonary gradient is imperative to maintain cardiac output. The ideal agent would be one that raises systemic vascular pressure while having a minimal effect on the pulmonary circulation.

One promising medication for treating hypotension in Fontan patients is vasopressin. One prior study evaluated the hemodynamic effect of vasopressin in pediatric patients with pulmonary hypertension. Compared to other vasopressor agents (phenylephrine, epinephrine), vasopressin increased systemic blood pressure with the least effect on pulmonary artery pressure. In a second study evaluating the use of vasopressin specifically for patients undergoing cardiac surgery for the creation of a Fontan, those who were treated with vasopressin as part of their postoperative management demonstrated lower transpulmonary gradients than those treated with placebo. Other studies have evaluated the use of vasopressin in Fontan patients for other clinical outcomes, such as decreasing postoperative chest tube output. On the basis of these studies, as well as our clinical experience managing these patients in the operating room, procedural suites, and in the intensive care unit, the investigator believes that vasopressin is not only safe but may be the preferred agent for this patient population.

Although vasopressin has been studied extensively in the context of sepsis, post cardiopulmonary bypass, and other vasoplegic disease states, the use of vasopressin has not yet been studied in the general population of patients who have Fontan physiology. The investigator hopes to demonstrate the efficacy of vasopressin as a medication specifically for these patients, as one that can elevate systemic blood pressure without compromising cardiac output or having a deleterious effect on the pulmonary vasculature.

ELIGIBILITY:
Inclusion Criteria:

1. All patients scheduled for cardiac catheterization at Lucile Packard Children's Hospital with Fontan circulation

Exclusion criteria:

1. Critical illness severe enough to preclude extended cardiac catheterization time
2. Patients already on vasopressin
3. Patients with pulmonary hypertension.
4. Patient not scheduled for cardiac catheterization at Lucile Packard Children's Hospital (LPCH).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change in systemic (aortic) blood pressure | Pre-dose, every 5 minutes post-dose for approximately 15 minutes (post-baseline values will be averaged)
Change in pulmonary artery pressure | Pre-dose, every 5 minutes post-dose for approximately 15 minutes (post-baseline values will be averaged)
Change in transpulmonary gradient | Pre-dose, every 5 minutes post-dose for approximately 15 minutes (post-baseline values will be averaged)
  Transpulmonary gradient = Mean pulmonary arterial pressure - left atrial pressure
PVR/SVR Ratio | Pre-dose, every 5 minutes post-dose for approximately 15 minutes (post-baseline values will be averaged)

CONTACTS AND LOCATIONS:
Overall Officials: Manchula Navaratnam, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamson GT, Yu J, Ramamoorthy C, Peng LF, Taylor A, Lennig M, Schmidt AR, Feinstein JA, Navaratnam M. Acute Hemodynamics in the Fontan Circulation: Open-Label Study of Vasopressin. Pediatr Crit Care Med. 2023 Nov 1;24(11):952-960. doi: 10.1097/PCC.0000000000003326. Epub 2023 Jul 18. PMID 37462430
- [Background] Siehr SL, Feinstein JA, Yang W, Peng LF, Ogawa MT, Ramamoorthy C. Hemodynamic Effects of Phenylephrine, Vasopressin, and Epinephrine in Children With Pulmonary Hypertension: A Pilot Study. Pediatr Crit Care Med. 2016 May;17(5):428-37. doi: 10.1097/PCC.0000000000000716. PMID 27144689
- [Background] Kumar TK, Kashyap P, Figueroa M, Zurakowski D, Allen J, Ballweg JA, Sathanandam S, Ali M, Knott-Craig CJ. Vasopressin After the Fontan Operation. World J Pediatr Congenit Heart Surg. 2016 Jan;7(1):43-8. doi: 10.1177/2150135115614574. PMID 26714993
- [Background] Bigelow AM, Ghanayem NS, Thompson NE, Scott JP, Cassidy LD, Woods KJ, Woods RK, Mitchell ME, Hraska V, Hoffman GM. Safety and Efficacy of Vasopressin After Fontan Completion: A Randomized Pilot Study. Ann Thorac Surg. 2019 Dec;108(6):1865-1874. doi: 10.1016/j.athoracsur.2019.06.053. Epub 2019 Aug 7. PMID 31400337